CLINICAL TRIAL: NCT00145665
Title: The Role of 3-Deoxy-3[18]Fluorothymidine Positron Emission Tomography (FLT-PET) in Proliferation of Colorectal Liver Metastases
Brief Title: The Role of Fluorothymidine Positron Emission Tomography (FLT-PET) in Proliferation of Colorectal Liver Metastases
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no accrual achieved
Sponsor: Radboud University Medical Center (Other)
Responsible Party: no sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: FLT-PET CRC-LM
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2007-02

CONDITIONS: Colorectal Neoplasms; Liver Neoplasms
Keywords: FLT-PET; colorectal liver metastases; proliferation; proliferation markers; recurrence
MeSH Terms: conditions — Colorectal Neoplasms; Liver Neoplasms; Recurrence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

INTERVENTIONS:
Procedure: FLT-PET scan — PET scan using FLT
  Other Names: [18F]-3'-fluoro-3'-deoxy-L-thymidine Positron emission tomography scan

SUMMARY:
The aim of the study is to obtain information on FLT used in a PET-scan as a marker for the proliferation of colorectal liver metastases, so that the risk of recurrence can be identified in a noninvasive way, concerning patients with resectable colorectal liver metastases.

The hypothesis of this study is that a higher uptake of FLT in the liver metastases has a good correlation with the proliferation rate of the metastases. This rate is related to the risk of recurrence.

DETAILED DESCRIPTION:
Aim of the Study:

Validation of FLT-PET as a proliferation marker for colorectal liver metastases, so that the risk of recurrence in patients with resected colorectal liver metastases can be assessed in a noninvasive method.

Study Design:

Validation study (n=40) to determine the correlation between quantitative FLT-PET (in this study determined before resection of the colorectal liver metastases) and the histologically determined proliferation index in the resected specimen of the metastases ('golden standard'). If correlation is established, the correlation between the proliferation and recurrence rate studied is also (n=80).

Study Population:

Patients with colorectal liver metastases.

Intervention:

FLT-PET scan

Scientific Basis of Study:

Several reports show that presence or absence of extrahepatic disease is a determining prognostic factor. Patients with extrahepatic disease are rarely suited for resection of the liver metastases. Recently several papers describe that the proliferation index of the liver metastases is another determining prognostic factor. Patients with a high proliferation factor have a worse prognosis. For both of these determining factors, it seems that PET diagnostics play an essential role and contribute to better selection of patients suitable for resection.

Diagnostics on Proliferation:

Seeing that the proliferation rate is preoperatively not determined without a biopsy (which is contraindicated due to dissemination), all patients with colorectal liver metastases (with no signs of extrahepatic deposits) are resected, without knowledge of the proliferation. FLT is a marker that visualizes proliferation and thus seems an ideal candidate to determine the proliferation rate in a noninvasive method. As of yet no validation studies of FLT-PET in colorectal liver metastases have been described.

Evaluation:

Quantitative histologic data are correlated with the quantitative FLT-PET data. If the correlation is higher that 0.85, this correlation is established. If this correlation is found, the inclusion of patients will be extended from 40 to 80 patients, seeing that this will give us the opportunity to correlate clinical data with the histological data. (alpha = 0.05, one-sided, beta = 0.90, assuming that an acceptable difference in sensitivity between both tests is 0 and an unacceptable difference is 0.02). If this correlation is significant, a new study will be proposed with the introduction of neoadjuvant chemotherapy, where the selection will be determined on basis of the proliferation rate.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal liver metastases deemed resectable on three-phase computed tomography (CT)-scan of the liver
* No evidence of extrahepatic disease on CT chest and abdomen and possible fluorodeoxyglucose (FDG)-PET (if part of surgical work-up)
* No evidence of local recurrence or second primary colorectal tumor on colonoscopy or colonography
* Primary colorectal tumor radically removed
* Informed consent

Exclusion Criteria:

* Pregnancy
* Recent chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
correlation FLT-uptake in colorectal liver metastases and the histologically determined proliferation

SECONDARY OUTCOMES:
correlation FLT and recurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: Bastiaan Wiering, MD, Principal Investigator — Radboud University Medical Center; Theo MJ Ruers, MD, PhD, Principal Investigator — Radboud University Medical Center; Wim JG Oyen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Fong Y, Cohen AM, Fortner JG, Enker WE, Turnbull AD, Coit DG, Marrero AM, Prasad M, Blumgart LH, Brennan MF. Liver resection for colorectal metastases. J Clin Oncol. 1997 Mar;15(3):938-46. doi: 10.1200/JCO.1997.15.3.938. PMID 9060531
- [Background] Hughes KS, Rosenstein RB, Songhorabodi S, Adson MA, Ilstrup DM, Fortner JG, Maclean BJ, Foster JH, Daly JM, Fitzherbert D, et al. Resection of the liver for colorectal carcinoma metastases. A multi-institutional study of long-term survivors. Dis Colon Rectum. 1988 Jan;31(1):1-4. doi: 10.1007/BF02552560. PMID 3366020
- [Background] Gibbs JF, Weber TK, Rodriguez-Bigas MA, Driscoll DL, Petrelli NJ. Intraoperative determinants of unresectability for patients with colorectal hepatic metastases. Cancer. 1998 Apr 1;82(7):1244-9. doi: 10.1002/(sici)1097-0142(19980401)82:73.0.co;2-f. PMID 9529015
- [Background] Tullo A, D'Erchia AM, Honda K, Mitry RR, Kelly MD, Habib NA, Saccone C, Sbisa E. Characterization of p53 mutations in colorectal liver metastases and correlation with clinical parameters. Clin Cancer Res. 1999 Nov;5(11):3523-8. PMID 10589767
- [Background] Buck AK, Schirrmeister H, Hetzel M, Von Der Heide M, Halter G, Glatting G, Mattfeldt T, Liewald F, Reske SN, Neumaier B. 3-deoxy-3-[(18)F]fluorothymidine-positron emission tomography for noninvasive assessment of proliferation in pulmonary nodules. Cancer Res. 2002 Jun 15;62(12):3331-4. PMID 12067968
- [Background] Buck AK, Halter G, Schirrmeister H, Kotzerke J, Wurziger I, Glatting G, Mattfeldt T, Neumaier B, Reske SN, Hetzel M. Imaging proliferation in lung tumors with PET: 18F-FLT versus 18F-FDG. J Nucl Med. 2003 Sep;44(9):1426-31. PMID 12960187
- [Background] Francis DL, Visvikis D, Costa DC, Arulampalam TH, Townsend C, Luthra SK, Taylor I, Ell PJ. Potential impact of [18F]3'-deoxy-3'-fluorothymidine versus [18F]fluoro-2-deoxy-D-glucose in positron emission tomography for colorectal cancer. Eur J Nucl Med Mol Imaging. 2003 Jul;30(7):988-94. doi: 10.1007/s00259-003-1187-0. Epub 2003 May 9. PMID 12739071
- [Background] Vesselle H, Grierson J, Peterson LM, Muzi M, Mankoff DA, Krohn KA. 18F-Fluorothymidine radiation dosimetry in human PET imaging studies. J Nucl Med. 2003 Sep;44(9):1482-8. PMID 12960196
- [Background] Rodgers MS, Collinson R, Desai S, Stubbs RS, McCall JL. Risk of dissemination with biopsy of colorectal liver metastases. Dis Colon Rectum. 2003 Apr;46(4):454-8; discussion 458-9. doi: 10.1007/s10350-004-6581-6. PMID 12682536